CLINICAL TRIAL: NCT05271994
Title: Fesibility of EUS-guided Gallbladder Drainage With a New-type of Electrocautery LAMS in the Treatment of Malignant Distal Biliary Obstruction
Acronym: DC LAMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas Mater Domini (Other)
Responsible Party: Sponsor
Other Study IDs: 01-2022
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Distal Malignant Biliary Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoscopic biliary drainage: Patients with distal malignant biliary obstruction, who need endoscopic biliary drainage
  Interventions: Procedure: endoscopic biliary drainage

INTERVENTIONS:
Procedure: endoscopic biliary drainage — endoscopic biliary drainage

SUMMARY:
Distal malignant biliary obstruction results from different types of tumors including pancreatic cancer, biliary tract cancer (BTC), gallbladder cancer, and metastasis, which can lead to obstructive jaundice. Endoscopic retrograde cholangiopancreatography (ERCP) represents the gold standard for jaundice palliation in this setting of patients. However, surgically altered anatomy (i.e., Whipple intervention, Roux-en-Y gastric bypass, Billroth II surgery), periampullary diverticula, gastric outlet obstruction, and malignant obstruction of the lumen determine the failure of the procedure in about 5-10% of cases, requiring alternative methods of decompression. Percutaneous transhepatic biliary drainage (PTBD) and surgical bypass are well established alternatives in these patients, but associated with increased morbidity, longer length of hospital stays and higher costs, and patient discomfort.

In 2001 Giovannini et al. described the first EUS guided biliary drainage (EUS-BD) through a transduodenal access with a needle knife. Subsequently, EUS-BD has considerably evolved thanks to the development of dedicated devices such as lumen apposing metal stents (LAMS), specifically designed for endoscopic ultrasound procedures. LAMS are made up of braided nitinol, that is fully covered with silicone to prevent tissue ingrowth, with wide flanges on both ends to provide anchorage.

Recently, LAMS have been incorporated into a delivery system with an electrocautery mounted on the tip (Hot Axios; Boston Scientific Corp.), which allows the device to be used directly to penetrate the target structure without the need to utilize a 19G needle, a guidewire, and a cystotome for prior dilation. This has been described for drainage of peri-pancreatic fluid collections, common bile duct (CBD), gallbladder, and for creation of gastro-jejuno anastomosis. The biliary drainage procedure performed with LAMS is a one step procedure that requires less or no need for accessory exchange and becomes faster, thus potentially decreasing the risk of complications.

The procedure has been described as safe and effective with a technical success of 98.2 %, clinical success of 96.4 %, and low rate of complications 7 % (duodenal perforations, bleeding and transient cholangitis) [6]. A systematic review and meta-analyses showed clinical and technical success rates of 87% and 95% respectively [7]. Currently, the EUS-BD is indicated as a rescue therapy for jaundice palliation after ERCP failure. Actually, only a retrospective series is published in literature about the gallbladder (GB) drainage in patients with malignant biliary obstruction (MBO), demonstrating the feasibility of gallbladder drainage to relieve malignant distal bile duct obstruction in patients with failed ERCP. No data are actually reported, especially in a prospective way, about the GB drainage as first intention in patients with MBO.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients with distal malignant biliary obstruction
* Gallbladder in place and accessible by EUS from the duodenum or from the stomach for the drainage
* Agree to receive follow up phone calls
* Able to provide written informed consent

Exclusion Criteria:

* Coagulation and/or platelets hereditary disorders and/or INR>1.5, PLT<50,000
* Use of anticoagulants that cannot be discontinued
* Pregnant women
* Inability to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational multicentric prospective study. Data from consecutive patients with jaundice caused by distal malignant biliary obstruction will be evaluated and, if eligible and agreed to participate, will be recorded in an electronic register. Patients will be followed until death or for at least 6 months (phone call at 1, 3 and 6 months).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Technical success | 2 years
  The rate of successful LAMS placement in the gallbladder
Clinical success | 2 years
  Decrease of the total bilirubin levels > 10% at 24 hours after procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas-Mater Domini, Castellanza, Italy

IPD SHARING:
Plan to Share IPD: No